CLINICAL TRIAL: NCT07258615
Title: Longitudinal Ultrasound Assessment of Diaphragmatic and Respiratory Muscle Function Following Respiratory Muscle Training in Frail Older Adults: A Randomized, Double-Blind, Sham-Controlled Trial
Brief Title: Longitudinal Ultrasound Assessment of Diaphragmatic and Respiratory Muscle Function Following Respiratory Muscle Training in Frail Older Adults
Acronym: IMT-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFV-IMT1
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Frailty Syndrome; Respiratory Muscle Weakness; Age-Related Frailty; Geriatric Health
Keywords: Inspiratory Muscle Training; Diaphragm Ultrasound; Older Adults
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training (Experimental): Participants perform an 8-week inspiratory muscle training program using a threshold device (PowerBreathe). Training consists of 30 inspirations, once daily, 5 days per week. The initial load is set at 50% of each participant's maximal inspiratory pressure (MIP) and is increased weekly by 5 cmH₂O up to 80% of MIP. All sessions are supervised by healthcare professionals, with continuous monitoring of oxygen saturation and heart rate.
  Interventions: Device: Inspiratory Muscle Training
- Inspiratory Muscle Training (Sham) (Sham Comparator): Participants follow the same 8-week training schedule using the threshold device (PowerBreathe), but with a constant load of 15% of maximal inspiratory pressure (MIP) and no weekly progression. Training consists of 30 inspirations, once daily, 5 days per week. The procedure mimics the experimental intervention but provides minimal physiological stimulus. All sessions are supervised, with monitoring of oxygen saturation and heart rate.
  Interventions: Device: Sham Inspiratory Muscle Training

INTERVENTIONS:
Device: Inspiratory Muscle Training — Participants perform 30 breaths once daily, 5 days per week for 8 weeks using a threshold inspiratory muscle training device. The load begins at 50% of maximal inspiratory pressure (MIP) and increases by 5 cmH₂O weekly up to 80% of MIP. Sessions are supervised and oxygen saturation and heart rate are monitored.
  Arms: Inspiratory Muscle Training
Device: Sham Inspiratory Muscle Training — Participants use the same device and schedule as the experimental group (30 breaths once daily, 5 days per week for 8 weeks) but with a constant load of 15% of maximal inspiratory pressure (MIP), with no weekly progression. This mimics the procedure while providing minimal physiological stimulus. Supervision and monitoring are identical to the experimental arm.
  Arms: Inspiratory Muscle Training (Sham)

SUMMARY:
This study aims to evaluate the effects of an 8-week inspiratory muscle training program on diaphragmatic and respiratory muscle function in frail older adults aged 80 years and above. Frailty is associated with reduced physical capacity, impaired respiratory performance, and a higher risk of disability. Inspiratory muscle training is a simple, low-cost intervention that may improve breathing function, strength, and overall health in very old adults, but evidence in this age group remains limited.

Participants will be randomly assigned to one of two groups: a high-load inspiratory muscle training group or a low-load sham training group. Both groups will use a threshold device and perform 30 breaths once per day, five days per week, for eight weeks. The experimental group will train with progressively increasing resistance (50% to 80% of maximal inspiratory pressure), while the sham group will use a minimal and non-progressive load (15% of maximal inspiratory pressure). All sessions will be supervised and monitored for safety.

The main goal of the study is to determine whether inspiratory muscle training improves maximal inspiratory pressure (MIP), an established measure of global inspiratory muscle strength. Secondary outcomes include ultrasound-based assessments of diaphragmatic structure and function, such as diaphragm thickness, contractile fraction, diaphragmatic excursion, inspiratory time, and inspiratory velocity during deep breathing and sniff maneuvers. These measurements will help clarify the physiological adaptations produced by inspiratory muscle training in this population.

Assessments will be performed before the intervention, immediately after the 8-week program, and again at one and three months after the end of the intervention to examine both immediate and short-term effects. This study may contribute valuable evidence regarding the safety, feasibility, and clinical benefits of inspiratory muscle training in frail very old adults, supporting its potential implementation in rehabilitation and geriatric care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 80 years or older.
* Clinical diagnosis of frailty, defined by a Short Physical Performance Battery (SPPB) score < 9.
* Ability to stand and walk with or without assistive devices.
* Ability to understand and follow instructions for inspiratory muscle training.
* Stable medical condition for at least 3 months prior to enrollment.
* Capacity to provide informed consent or availability of a legal representative.

Exclusion Criteria:

* Acute or unstable cardiovascular, respiratory, or metabolic conditions.
* Severe cognitive impairment that prevents understanding the procedures.
* Diagnosis of neuromuscular diseases affecting respiratory muscles (e.g., ALS, myopathies).
* Severe or uncontrolled hypertension (≥180/110 mmHg).
* Recent thoracic or abdominal surgery (<3 months).
* Severe musculoskeletal disorders limiting participation in training.
* History of recurrent syncope, severe dizziness, or intolerance to respiratory maneuvers.
* Any condition judged by the research team to compromise safety or participation.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure (MIP) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Maximal Inspiratory Pressure (MIP) will be measured using a calibrated handheld manometer following standardized respiratory assessment guidelines. Participants will be instructed to perform a maximal inspiratory effort from residual volume through the mouthpiece with their nose occluded. At least three maneuvers will be recorded, ensuring less than 10% variability between attempts. The highest reproducible value (cmH₂O) will be used for analysis. This measure reflects global inspiratory muscle strength and is widely validated in older and frail populations.

SECONDARY OUTCOMES:
Diaphragm Thickness at End-Expiration (DTE) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Diaphragm thickness at end-expiration will be measured using 2D ultrasound at the zone of apposition. Three measurements will be obtained and averaged. This variable reflects diaphragm muscle thickness at rest.
Diaphragm Thickness at End-Inspiration (DTi) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Diaphragm thickness at end-inspiration will be measured using 2D ultrasound during a maximal inspiratory effort. Three measurements will be averaged. This variable reflects diaphragm contraction thickness.
Diaphragm Thickening Fraction (DTF) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  The diaphragm thickening fraction will be calculated as:
  Diaphragm Thickening Fraction (DTF) = [(Diaphragm Thickness at End-Inspiration (DTi) - Diaphragm Thickness at End-Expiration (DTE)) / DTE] × 100.
  This percentage reflects diaphragm contractile capacity.
Diaphragmatic Excursion During Deep Breathing (DMDB) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Diaphragmatic excursion during deep breathing will be assessed with M-mode ultrasound during a maximal inspiratory maneuver. The average of three reproducible measurements will be used to quantify the cranio-caudal diaphragm displacement.
Inspiratory Time During Deep Breathing (DTDB) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Inspiratory time during deep breathing will be measured from the M-mode tracing as the time from the onset of diaphragm movement to its maximal excursion. This reflects the temporal characteristics of deep inspiration.
Inspiratory Velocity During Deep Breathing (DVDB) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Inspiratory velocity will be calculated by dividing diaphragmatic excursion (DMDB) by inspiratory time (DTDB), providing an estimate of average inspiratory velocity.
Diaphragmatic Excursion During Sniff Maneuver (DMVS) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Diaphragmatic excursion during a voluntary sniff will be measured with M-mode ultrasound during a rapid, forced nasal inspiration. The average of three reproducible efforts will be used to quantify rapid diaphragm displacement.
Inspiratory Time During Sniff Maneuver (DTVS) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Inspiratory time during the sniff maneuver will be measured from the start of diaphragm movement to its peak excursion on the M-mode tracing.
Inspiratory Velocity During Sniff Maneuver (DVVS) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Inspiratory velocity during sniff will be calculated by dividing sniff excursion by the corresponding inspiratory time, reflecting rapid contractile performance.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Sánchez-Infante, PhD, PT, Principal Investigator — Universidad Francisco de Vitoria

IPD SHARING:
Plan to Share IPD: Undecided
At this time, it is unclear whether individual participant data (IPD) will be shared. Data sharing will depend on institutional policies, ethical approvals, participant privacy considerations, and the feasibility of preparing de-identified datasets. A final decision will be made once data collection and analysis are completed.